CLINICAL TRIAL: NCT05617131
Title: Feasibility Study of the Implementation of a Cell Phone Application to Help Adolescents and Young Adults in Their Therapeutic and Educational Journey
Brief Title: Cell Phone Application to Help Adolescents and Young Adults in Their Therapeutic and Educational Journey
Acronym: OnKO-TnT-1-0
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7599
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Cancer
Keywords: Solid cancer; Liquid cancer; Connected health tools; OnKO-TnT digital application
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
About 2000 cancers/year in France are diagnosed in Adolescents and Young Adults (15-25 years old, AYA). The cancer plans and the INCA recommend support during and after cancer, taking into account both medical and psychosocial specificities related to age (supportive care, school learning/training and professional integration, fertility preservation, therapeutic education, addictology, sexology...). The care offered is often heterogeneous for these AYAs in transition between the pediatric and adult worlds. They may be cared for either in pediatric oncology units or in adult structures. In this context, an AYA team has been developed in the Strasbourg center, led by a Nurse Coordinator (IDEC), social workers, psychologists and doctors. Thus, the young patients and their relatives are accompanied by professionals during their therapeutic care. In spite of this global care and closer to the patient, it is still necessary to find connected health tools for these AYA.

DETAILED DESCRIPTION:
In this context, the Strasbourg team has initiated the development of a digital application compatible for any cell phone OnKO-Tips &Tricks meeting these criteria of necessity. The application is currently in its final phase and requires validation by patients through a feasibility study that will last 6 months. Thus, all patients currently followed or newly diagnosed with liquid or solid cancer and aged between 15 and 25 years old will be included and will have the opportunity to test the application, its practicality as well as its current use and in particular its expected benefits for an optimization of our ETP program.

ELIGIBILITY:
Inclusion criteria:

* Subject whose age is ≥ 15 years and ≤ 25 years
* Subject diagnosed at the Strasbourg center (HUS and ICANS) with solid or liquid cancer
* Subject followed in the Strasbourg center (HUS and ICANS)
* Subject (or his/her legal representatives) having given his/her (their) agreement to participate in the evaluation survey of the OnKO-TnT digital application
* Subject agreeing to complete all satisfaction questionnaires
* The subject understands, speaks and writes French fluently
* Subject having a cell phone capable of downloading the application (developed for any type of cell phone)

Criteria for non-inclusion :

* Opposition of the subject (or the holders of parental authority) to participate in the satisfaction survey
* Subject under legal protection
* Subject under guardianship or curatorship

Ages: 15 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Subject, whose age is ≥ 15 years and ≤ 25 years, diagnosed at the Strasbourg center (HUS and ICANS) with solid or liquid cancer
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Collection of the global score of the MAUQ questionnaire (item 1 to 21), filled in by the patients after 6 months of use of the OnKO-TnT application | after 6 months of use of the OnKO-TnT application
  MAUQ questionnaire of 21 items with a score ranging from 1 to 7. Score 7 means a better result

CONTACTS AND LOCATIONS:
Locations (1):
- Service Pédiatrie Onco-hématologie - Pédiatrie III - CHU de Strasbourg - France, Strasbourg, France